CLINICAL TRIAL: NCT01903759
Title: Kinetics of Inflammation Markers in Maternal Plasma (Interleukins, Matrix Metalloproteinases -MMP): Study of the Correlation With the Diagnosis of Chorioamnionitis in Women Hospitalized for Spontaneous Rupture of the Fetal Membranes (SPROM) Before 34 Weeks of Amenorrhea (WA) With no Modification in the Usual Therapy.
Brief Title: Kinetics of Inflammation Markers in Maternal Plasma: Study of the Correlation With the Diagnosis of Chorioamnionitis in Women Hospitalized for Spontaneous Rupture of the Fetal Membranes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Sagot PHRC IR 2006
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Patients With Spontaneous Rupture of the Fetal Membranes
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with spontaneous rupture of the fetal membranes (Other)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
The principal aim of this study is to help obstetricians to diagnose chorioamniotic infection early, in cases of premature rupture of the fetal membranes before 34 WA, by proposing earlier and more specific markers of infection than FBC and CRP. The aim is to reduce vital and functional risk of acute chorioamnionitis for the mother, the fetus or the newborn,.

If the kinetics profile of one or several markers correlates strongly with the diagnosis of chorioamnionitis, it could be used in clinical practice, possibly in the context of another clinical study.

The results of the study presented here are destined to be published in obstetrics journals.

ELIGIBILITY:
Inclusion Criteria:

* Term between 24 and 34 WA
* Spontaneous rupture of the fetal membranes
* Singleton pregnancy
* Age > 18 years

Exclusion Criteria:

* Delivery within the hour following admission
* Hospitalisation before 24 WA or after 34 WA
* Hemorrhagic placenta previa or retroplacental hematoma, known auto-immune or inflammatory disease
* Infection with human immunodeficiency virus (HIV)
* Refusal to provide consent.
* Patients provided for in articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code (e.g.: minors, adults under guardianship, etc…)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
determination of plasma cytokines | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France